CLINICAL TRIAL: NCT03862664
Title: Respiratory Complications Among Living Liver-donors: a Single Center Observational Retrospective Study
Brief Title: Respiratory Complications Among Living Liver-donors
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohammed Sayed Shorbagy, Lecturer of Anesthesia, Ain Shams University
Other Study IDs: FAMSU R37/2018
Record Dates: First submitted 2019-02-25; First posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Complication of Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Collection of data — The investigators will retrieve retrospectively the medical record of donors who underwent hepatic lobectomy for liver transplantation

SUMMARY:
Recently, there are increasing reports about pulmonary complications within living liver donors postoperatively. In this retrospective study, the investigators will highlight the risk factors and incidence of pulmonary complication among living liver-donors in our center.

ELIGIBILITY:
Inclusion Criteria:

* Excellent general physical and mental condition,
* Free of chronic disease or
* Previous major abdominal surgery,
* Body mass index (BMI) <28,
* ABO blood group identical to recipients and
* Negative for hepatitis B, C and human immunodeficiency viruses (HIV).

Exclusion Criteria:

* ASA physical status> II,
* BMI>28,
* Psychiatric or mental retardation,
* pregnant and nursing women or
* Patients with significant laboratory abnormalities

Ages: 20 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Donors who underwent hepatic lobectomy for liver transplantation
Sampling Method: Probability Sample
Enrollment: 124 (Estimated)
Dates: Start 2019-02-06 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
The number of participants with postoperative respiratory complications | an average period of 3 year
  Respiratory complications as pulmonary embolism, pleural effusion, pneumothorax, pneumonia, atelectasis, acute lung injury (ALI), acute respiratory distress syndrome (ARDS), and transfusion-related acute lung injury (TRALI) will be considered when they are clinically evident.

SECONDARY OUTCOMES:
The average of ICU stay among patients | an average period of 3 year
  It is defined as time period from entry to ICU till discharge to the ward
The average of hospital stay among patients | an average period of 3 year
  It is defined as time period elapsed from discharge to the ward till leaving the hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided